CLINICAL TRIAL: NCT02356835
Title: A Pivotal Study of the Use of Nitric Oxide / Plasma Therapy as Produced by the APT001 Plasma / Nitric Oxide Generator in Adult Subjects With a Diabetic Foot Ulcer
Brief Title: APT001 Plasma/NO Generator to Treat Diabetic Foot Ulcer in Adults
Acronym: APT-14-002
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Origin Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APT-14-002
Record Dates: First submitted 2015-02-03; First posted 2015-02-05 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- APT001 (Experimental): The APT001 is a medical device that generates a plasma flow containing nitric oxide intended to be applied topically to wound sites. The nitric oxide / plasma flow will be directed at the wound site and surrounding skin at a distance of 11.5 to 15 centimeters from the skin surface. Dose will be 10 seconds / cm2 wound surface area. Administration of the therapy will include a 2 cm border around the defined edges of the wound site.
  Interventions: Device: APT001
- SHAM (Sham Comparator): Treatment with a sham device to deliver non-medicated, heated room air to the wound in the same manner and dose as the active treatment device.
  Interventions: Device: SHAM

INTERVENTIONS:
Device: APT001 — APT001, is a portable device that uses plasma energy to deliver nitric oxide to the tissues.
  Other Names: APT001 Plasma/Nitric Oxide
  Arms: APT001
Device: SHAM — Portable device that uses warmed room air to mimic delivery of the APT001 treatment.
  Arms: SHAM

SUMMARY:
This is a 10-week, randomized, controlled study to evaluate the efficacy and safety of the APT001 plasma and nitric oxide treatment in subjects with a diabetic foot ulcer.

DETAILED DESCRIPTION:
Approximately 80 subjects will be randomized by computer to receive equally either sham therapy or plasma / nitric oxide treatments topically. The nitric oxide / plasma treatment will be delivered from 11.5 to 15 centimeters from the wound surface for 10 seconds per cm2 of wound size. Subjects will be evaluated for efficacy and safety on a regular basis with clinical observations. The wounds of both groups will be treated with sharp debridement as determined by the site Investigator. A collagen dressing, a non-adherent dressing, and an absorptive dressing will be applied to the wound after either the study therapy or the sham therapy.

For an initial safety evaluation in patients with DFU, the first ten patients randomized will be limited to wound size of 7 cm2 or less and their wounds will be assessed 2-4 days after each treatment session. Following completion of the final assessment in these 10 patients, data will be submitted to FDA for review and approval before opening the enrolment for the remaining patients.

ELIGIBILITY:
Inclusion Criteria:

* 19 to 80 years of age
* Type 1 or 2 diabetes with hemoglobin A1c less than 12%
* ABI ≥ 0.7, palpable pulses and/or biphasic waveform study with Doppler
* Wound size ≥ 1cm2 and ≤ 30cm2 (the first 10 patients enrolled will be limited to a wound size of 7 cm2 or less)

Exclusion Criteria:

* Have a significant concomitant illness that would adversely affect participation in the study or affect the healing of the wound
* Have a severe infection in the ulcer including the presence of an abscess, cellulitis extending > 2 cm beyond the ulcer margin, or osteomyelitis
* Have involvement of deeper tissues including bone or tendon
* Be currently receiving steroid medications, chemotherapy, or other medications that might affect healing of the wound
* Have received topical or systemic antimicrobial therapy within 48 hours of screening
* Have a malignancy other than skin cancer currently being treated
* Have substance abuse issues within the 6 months prior to screening
* Is a woman who is pregnant or breast feeding
* Has been treated with another investigational product within 30 days of screening
* Has been treated with tissue engineered skin or a biological therapy within 30 days of screening

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percent change in total wound size | Baseline to end of Week 10
  Change in total wound size using dimensional measurements of the wound and using the Aranz SilhouetteStar + SilhouetteConnect wound assessment device from Baseline to Week 10.

SECONDARY OUTCOMES:
Change in bacterial load | Baseline to end of Week 5
  Clearance of wound infection based on clinical observation and wound biopsy cultures.
Wound pain | Baseline to end of Week 10
  Wound pain measured by a standard wound pain scale completed at each visit prior to treatment or any study procedures.

CONTACTS AND LOCATIONS:
Overall Officials: David R Dantzker, MD, Study Director — Origin Inc.; Terry A Treadwell, MD, Principal Investigator — Institute for Advanced Wound Care Baptist Health
Locations (3):
- United States (3):
  - Baptist Health Institute for Advanced Wound Care, Montgomery, Alabama
  - Limb Preservation Platform, Inc., Fresno, California
  - New York College of Podiatric Medicine, New York, New York